CLINICAL TRIAL: NCT01077050
Title: SciBase International Melanoma Pivotal Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SciBase AB (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: SIMPS
Record Dates: First submitted 2010-02-25; First posted 2010-02-26 (Estimated); Results first posted 2013-12-30 (Estimated); Last update posted 2013-12-30 (Estimated); Status verified 2013-11

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (1):
- SciBase III (Other): Subjects with suspected malignant melanoma or lesions designated for total excision were included into the study. To ensure no selection bias, all eligible lesions from a subject were included into the study. All study eligible skin lesion(s) were examined with the investigational device, photographed and removed by an excisional biopsy.
  Interventions: Device: SciBase III Electrical Impedance Spectrometer

INTERVENTIONS:
Device: SciBase III Electrical Impedance Spectrometer — SciBase III Electrical Impedance Spectrometer is based on Electrical Impedance Spectroscopy (EIS). EIS is a measure of the overall resistance within a skin tissue, at alternating currents of various frequencies. Enrolled subject will undergo skin measurements with SciBase III Electrical Impedance Spectrometer. The relevant skin lesion(s) will be excised and diagnosed as per routine treatment.

SUMMARY:
The purpose of this clinical investigation was to determine the safety and effectiveness of the SciBase III device (Test) designed to help distinguish between malignant melanoma and benign lesions, using electrical impedance spectroscopy (EIS) relative to the histological gold standard (Reference).

The purpose of the study is to collect data to support a Pre-market Application(PMA) to obtain Food and Drug Administration(FDA) approval to market the SciBase III Electrical Impedance Spectrometer.

ELIGIBILITY:
Inclusion Criteria

For inclusion in the study, all subjects had to fulfill all of the following criteria:

* Men or women of any ethnic group aged ≥18 years
* Primary lesions (i.e., not metastases or recurrent lesions) that the physicians choose to excise.
* Lesion ≥ 2 mm in diameter and ≤ 20 mm in diameter
* In subjects with multiple skin lesions, all lesions destined for excision must be identified for purposes of study participation. Note: a subject may only be entered into the study once.
* The subject is willing and able to read, understand and sign the study specific informed consent form.

Exclusion Criteria:

Subjects were excluded from the study if they fulfilled any of the following criteria:

* Skin surface not measurable, e.g. lesion on a stalk
* Skin surface not accessible, e.g. inside ears, under nails
* Lesion located on acral skin, e.g. sole or palms.
* Lesion located on areas of scars, crusts, psoriasis, eczema or similar skin conditions.
* Lesion on hair-covered areas, e.g. scalp, beards, moustaches or whiskers.
* Lesion located on genitalia.
* Lesion located in an area that has been previously biopsied or subjected to any kind of surgical intervention or traumatized.
* Lesion located on mucosal surfaces.
* Skin is not intact (measurement area) e.g. bleeding or with clinical noticeable ulceration.
* Lesion with foreign matter, e.g. tattoo, splinter
* Lesion and/or reference located on acute sunburn.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1951 (Actual)
Dates: Start 2010-04; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik H Birgersson, PhD, Study Director — SciBase and Karolinska Institutet
Locations (2):
- University of Arizona, Tucson, Arizona, United States
- Sahlgrenska University Hospital, Gothenburg, Sweden

REFERENCES:
- [Background] Aberg P, Nicander I, Holmgren U, Geladi P, Ollmar S. Assessment of skin lesions and skin cancer using simple electrical impedance indices. Skin Res Technol. 2003 Aug;9(3):257-61. doi: 10.1034/j.1600-0846.2003.00017.x. PMID 12877688
- [Background] Aberg P, Nicander I, Hansson J, Geladi P, Holmgren U, Ollmar S. Skin cancer identification using multifrequency electrical impedance--a potential screening tool. IEEE Trans Biomed Eng. 2004 Dec;51(12):2097-102. doi: 10.1109/TBME.2004.836523. PMID 15605856

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted at five (5) US investigational sites and at seventeen (17) European investigational sites.
  Recruitment period 2010-2011. In 2012 the last histological analysis was performed.
Pre-assignment Details: Potential study subjects were screened according to the inclusion/exclusion criteria. All study eligible skin lesion(s) were then examined with the investigational device, photographed and removed by an excisional biopsy.
Period: Overall Study
Arm/Group | Only One Arm in the Study, Thus Not Applicable.
Started | 1951
Completed | 1942
Not Completed | 9
Not completed — Subjects signed ICF could not be located | 1
Not completed — Screen failure | 8

BASELINE CHARACTERISTICS:
Population: All study eligible skin lesion(s) were examined with the investigational device, photographed and removed by an excisional biopsy.
Groups:
- Biopsied Skin Lesions: Lesions for which clinical management was prospectively determined to be biopsy of the lesion in toto
Arm/Group | Biopsied Skin Lesions
Number analyzed (Participants) | 1942
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1499
  >=65 years | 443
Age Continuous [Mean (Standard Deviation); unit: years] | 49.8 (16.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1013
  Male | 929
Region of Enrollment [Number; unit: participants]
  United States | 458
  Europe | 1484

OUTCOME MEASURES:

1. Primary Outcome: SciBase Sensitivity and Specificity
Description: This study has two co-primary objectives, aiming to demonstrate the accuracy of SciBase device:
  1. Sensitivity ≥ 0.90 to detect Melanoma
  2. Sensitivity - (1-Specificity) > 0.00
  Sensitivity is the proportion of correctly identified cases of Melanoma. Specificity is the proportion of correctly identified cases of non-melanoma.
Time Frame: Post data lock
Population: Biopsied Skin Lesions
Measure: Mean (95% Confidence Interval); unit: Percentage of total lesions
Units Other Than Participants: Biopsied Skin Lesions
Arm/Group | Biopsied Skin Lesions
Number analyzed (Participants) | 1611
Number analyzed (Biopsied Skin Lesions) | 1943
Percentage of total lesions
  SciBase Sensitivity to melanoma | 96.6 [93.7 to 98.4]
  SciBase Specificity to non-melanoma | 31.4 [29.2 to 33.7]
Statistical Analysis 1: Comparison: Biopsied Skin Lesions; Test type: Superiority or Other; Clopper-Pearson 1-sided — The point estimate of the observed sensitivity that is based on generalized linear mixed model is equal to that calculated in the usual manner; Sensitivity to Melanoma = 96.6, 95% CI 1-sided [lower limit 94.2]
Statistical Analysis 2: Comparison: Biopsied Skin Lesions; Test type: Superiority or Other; Clopper-Pearson 2-sided; Point estimate of the observed sensitivity for Basal Cell Carcinoma; Sensitivity to Basal Cell Carcinoma = 100, 95% CI 2-sided [92.6 to 100]
Statistical Analysis 3: Comparison: Biopsied Skin Lesions; Test type: Superiority or Other; Clopper-Pearson 2-sided; Point estimate of the observed sensitivity for squamous cell carcinoma; Observed sensitivity for squamous cell c = 93.3, 95% CI 2-sided [68.1 to 99.8]
Statistical Analysis 4: Comparison: Biopsied Skin Lesions; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Note that calculating odds ratio adjusting for subjects having multiple lesions, yields similar result; Odds Ratio (OR) = 13.0, 95% CI 2-sided [6.6 to 25.5]

2. Secondary Outcome: Sensitivity and Specificity
Description: Secondary confirmatory objective included two co-secondary endpoints that were defined similarly to the co-primary endpoints, but used the Secondary definition of dichotomous reference diagnosis.
  Positive Reference Diagnosis: Melanoma, Squamous Cell Carcinoma, Basal Cell Carcinoma, Severe Dysplastic Nevus (High grade dysplasia)
  Negative Reference Diagnosis: All other skin lesions.
Time Frame: Post data lock
Reporting Status: Not Posted, anticipated posting 2013-08

ADVERSE EVENTS:
Time Frame: A post-procedure follow up, either by a telephone or investigational site visit, was to be conducted at 7 (seven) +/- 3 (three) days from the SciBase III evaluation, at which time the subject were to be evaluated for any adverse events.
Description: The Safety analysis population includes all subjects for whom there was any contact with subject's skin and the SciBase III investigational device. Therefore the number of subjects included in the safety analysis deviates from both the total number of enrolled and eligible subjects.
Groups:
- Biopsied Skin Lesions: Any adverse advent that occured on a skin/lesion site for whom there had been any contact between the subject's skin and investigational device (SciBase III).
  Note that multiple adverse event occured on some subjects. In total 36 Adverse Events were reported on 28 subjects.
Arm/Group | Biopsied Skin Lesions
Serious Adverse Events (participants affected / at risk) | 0/1915
Other Adverse Events (participants affected / at risk) | 28/1915
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Biopsied Skin Lesions (N=1915)
Experienced bleeding through the bandage after excision. (Skin and subcutaneous tissue disorders) | 2 (2)
Experienced a headache/migrane post SciBase measurements and surgical excision. (Nervous system disorders) | 4 (4)
Lesion started to bleed during examination/measurement (Skin and subcutaneous tissue disorders) | 6 (6)
Experience of slight pain from excision (Skin and subcutaneous tissue disorders) | 3 (3) — Experienced pain from the wound or excisional site.
Experience of slight pain/pin pricks from probe (Skin and subcutaneous tissue disorders) | 4 (4) — Experienced slight pain / pin pricks from the probe. Resolved once the probe was removed or measurements ended.
Experience of soreness/itch/tingling at excisional/measurement site (Skin and subcutaneous tissue disorders) | 5 (5)
Developed infection following excision (Skin and subcutaneous tissue disorders) | 4 (4)
Suffered from a cold (General disorders) | 1 (1) — Suffered from a cold for 3 days after the excision had been performed.
Neck and facial swelling after lymph node dissection (Blood and lymphatic system disorders) | 1 (1) — Suffered from neck and facial swelling 2 days after lymph node dissection surgery had been performed.
Experience nausea (General disorders) | 1 (1) — Experience nausea for 2 days post measurement and excision
Suffered from diarrhea (Gastrointestinal disorders) | 1 (1) — Suffered from diarrhea for two days after measurements and excision
Suture came out prematurely (General disorders) | 1 (1) — One suture came out prematurely.
Minimal brusing (Skin and subcutaneous tissue disorders) | 1 (1) — Experienced very minimal bruising appeared on the measurement site approximately 10 minutes after four attempts had been made to obtain a device reading.
Experienced sensation of fainting (General disorders) | 1 (1) — Became pale and felt faint immediately following the biopsy. The subject felt much better after lying down and was able to leave the clinic under his own power.
Experienced mild chest pain (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less